CLINICAL TRIAL: NCT01656863
Title: Oral Rehydration Therapy in Children With Mild to Moderate Dehydration
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 00-15-12 HYMC
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Parent; Attitudes
Keywords: Dehydration
MeSH Terms: conditions — Behavior; Dehydration | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Parents: Parents reporting to the emergency room with dehydrated children
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire

SUMMARY:
The purpose of this study is to determine parental attitudes towards oral rehydration therapy for children with mild to moderate dehydration.

ELIGIBILITY:
Inclusion Criteria:

* Parents of dehydrated children aged 0-18

Exclusion Criteria:

* Child with severe dehydration
* Child with chronic disease causing dehydration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents of children suffering dehydration reporting to pediatric emergency room
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel